CLINICAL TRIAL: NCT06398405
Title: Efficacy and Safety of Epigallocatechin-3-gallate, an Important Polyphenolic That Originates From Tea, in Patients With Esophageal Squamous Cancer: A Phase II Trial
Brief Title: A Phase II Clinical Study of Epigallocatechin-3-gallate in Patients With Esophageal Squamous Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, Deputy Chief Physician, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTEEC2024
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer; Dysphagia, Esophageal; Epigallocatechin Gallate
Keywords: Esophageal Cancer; Dysphagia, Esophageal; Epigallocatechin gallate
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders | interventions — epigallocatechin gallate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EGCG ARM (Experimental): Studies investigating EGCG (purity 95% by high-performance liquid chromatography, obtained from Zhejiang Ningbo HEP Biotech Co., Ltd.) utilized a concentration of 4400 umol/L dissolved in 0.9% saline solution, which is administered three times a day for 1 week. Freshly prepared each time, the EGCG was administered 10 minutes before meals. The repeated slow swallowing of 30 ml of the EGCG solution was essential to ensure sustained contact of the drug on the esophageal walls
  Interventions: Other: Epigallocatechin-3-gallate

INTERVENTIONS:
Other: Epigallocatechin-3-gallate — Epigallocatechin-3-gallate is administered in a solution with a concentration of 4400 umol/L

SUMMARY:
The investigators conduct this phase II study to evaluate safety and effectiveness of EGCG in patients with dysphagia. Swallowing-related dysphagia and pain scores were recorded using the numerical rating scale (NRS) daily . Barium meal radiography was utilized to measure the luminal size and the length of the lesion area both before and after a week of EGCG treatment. The scales are translated into Chinese and guides in Chinese are developed instructing how to use the scales and perform the assessments.

ELIGIBILITY:
Inclusion Criteria:

* confirmed pathological esophageal squamous cell carcinoma
* ≥18 years old
* the Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1
* no previous anti-tumor treatment
* no esophageal bleeding or fistula
* adequate hemocyte count, normal hepatic and renal functions
* Esophageal obstruction classified as grade 2 or grade 3 according to Stooler's dysphagia score

Exclusion Criteria:

* lactating or pregnant women
* known hypersensitivity or allergy to any kind green tea extract
* placement of small intestinal feeding tube or endoscopic stent treatment
* unable or refusing to take oral liquids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Choking symptom objective response rate | baseline and up to 7 days post-treatment
  Choking when swallowing was assessed by Stooler's dysphagia score (0-4, with 0 being none and 4 being completely unable to feed orally)
Pain symptom objective response rate | baseline and up to 7 days post-treatment
  Pain when swallowing was assessed by numerical rating scale (0-5, with 0 being none and 5 being worst pain imaginable)
Imaging objective response rate | Change from Baseline esophageal stenosis size at 7 days
  Response rate of esophageal stenosis was determined by X-ray barium meal examination and/or contrast-enhanced CT

SECONDARY OUTCOMES:
prealbumin change | baseline and up to 7 days post-treatment
  The prealbumin values were tested by biochemical analysis
Albumin change | baseline and up to 7 days post-treatment
  The albumin values were tested by biochemical analysis
Number of Participants with Adverse Events | baseline and up to 7 days post-treatment
  participants will be followed for the duration of EGCG treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China